CLINICAL TRIAL: NCT02782026
Title: Exhaled Breath Olfactory Signature of Pulmonary Arterial Hypertension Detected by an Artificial Nose: A Clinical Validation Study
Brief Title: Exhaled Breath Olfactory Signature of Pulmonary Arterial Hypertension
Acronym: SNOOPY2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Technion, Israel Institute of Technology (Other); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-01321-46
Record Dates: First submitted 2016-02-23; First posted 2016-05-25 (Estimated); Last update posted 2021-05-04 (Actual); Status verified 2016-12

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; early detection
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — Electronic Nose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- idiopathic PAH (Experimental): Exhaled Breath Olfactory Signature Detected by an Artificial Nose
  Interventions: Device: Exhaled Breath Olfactory Signature (Artificial Nose)
- heritable PAH with BMPR2 mutation (Experimental): Exhaled Breath Olfactory Signature Detected by an Artificial Nose
  Interventions: Device: Exhaled Breath Olfactory Signature (Artificial Nose)
- chronic thromboembolic PH (Experimental): Exhaled Breath Olfactory Signature Detected by an Artificial Nose
  Interventions: Device: Exhaled Breath Olfactory Signature (Artificial Nose)
- Controls (Experimental): Exhaled Breath Olfactory Signature Detected by an Artificial Nose
  Interventions: Device: Exhaled Breath Olfactory Signature (Artificial Nose)

INTERVENTIONS:
Device: Exhaled Breath Olfactory Signature (Artificial Nose)

SUMMARY:
In this prospective case-control study, the investigators will evaluate the diagnostic performance of a novel electronic nose (E-nose) for the detection of Pulmonary Arterial Hypertension (PAH). This study is designed to:

1. Assess the performance of the E-nose to discriminate controls from patients with PAH
2. Assess the performance of the E-nose to discriminate between different subtypes of pulmonary hypertension (PH), namely idiopathic PAH, heritable PAH with BMPR2 mutation and chronic thromboembolic PH
3. Assess the performance of the E-nose to discriminate controls from asymptomatic patients with PH who carry BMPR2 mutations.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension (PAH) is a progressive and rare severe disease (prevalence of 15-50 per million) due to obstruction of small pulmonary arteries, leading to an increase in pulmonary artery pressure with the ultimate consequence right heart failure. Despite recent advances in therapeutic care, there is no cure and most patients die or require lung transplantation within 5 years of diagnosis. Currently, right heart catheterisation is required to diagnose PAH and monitor response to treatment. Right heart catheterisation is an invasive test, and alternatives such as echocardiography have not yielded sufficient accuracy both for early diagnosis and disease monitoring. Currently, PAH is often diagnosed at an advanced stage of the disease. There is often a delay in diagnosis of several years between the first symptoms and the identification of the disease due to the non-specific nature of symptoms. Hence, there is the need to improve the time between the first signs and definitive diagnosis of the disease. Early diagnosis of PAH remains a challenge due to the low sensitivity and specificity of biomarkers available currently.

The main objective is to validate the results obtained in the previous preliminary proof of concept study - that PAH patients display a unique olfactory signature that can be detected by an artificial E- nose.

Secondary objectives are to investigate the ability of the E-nose to:

* Discriminate patients with idiopathic PAH from those with heritable PAH due to BMPR2 mutations
* Discriminate patients with chronic thromboembolic pulmonary hypertension (CTEPH) from healthy controls, and patients with idiopathic and/or heritable PAH.
* Detect development of PAH in BMPR2 mutation carriers
* Determine whether the olfactory signature can stratify subgroups of patients by correlating the olfactory signature to different biological and clinical parameters (hemodynamic measurements, NYHA class, duration of treatment, 6-minute walk distance, response to nitric oxide, BNP levels).

ELIGIBILITY:
Inclusion Criteria:

Patients group (Group A)

* Age 18 to 65 years inclusive
* Idiopathic or heritable PAH confirmed by right heart catheterization
* Affiliated to a social security (excluding AME)

Healthy control group (Group B)

* Age 18 to 65 years inclusive
* No known allergy
* No history of known pathology
* No chronic disease in active phase
* No history of respiratory illness
* Not genetically linked with the patient
* Affiliated to a social security (excluding AME)

At risk group (Group C)

* Age between 18 and 65 years old inclusive
* Subjects included in the protocol Delphi2 or Subject satisfying the inclusion and non-inclusion criteria of the DELPHI2 study
* Affiliated to a social security (excluding AME)

Patient group (Group D)

* Age between 18 and 65 years old inclusive
* Post-embolic HTP
* Affiliated to a social security scheme (excluding AME)

Exclusion Criteria:

Any patient/subject presenting :

* Connective tissue disease
* HIV infection
* Portal hypertension
* Congenital heart disease
* Asthma and other coexisting lung diseases
* Pregnant or breastfeeding woman
* Alcohol addiction (if consumption >3 glasses/day for men and >2 glasses/day for women)
* Smoking addiction (if consumption >5 cigarettes/day)
* Having had a CT scan in the week prior to the inclusion visit
* Subjects who have consumed coffee, alcohol, or a cigarette in less than 3 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2016-03-04 (Actual); Primary Completion 2018-08-28 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Volatile organic compounds in exhaled breath in patients of each group detected using sensor array on the basis of cross-reactive gold-nanoparticles coated with organic ligands. | Up to 4 hours
  The primary endpoint will be the ability of the E-nose to discriminate patients with PAH from healthy controls by their olfactory signature from the profile of volatile organic compounds in exhaled breath.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Humbert, MD,PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Bicêtre Hospital, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No